CLINICAL TRIAL: NCT06652282
Title: Effect of Pilates Exercise Versus Proprioceptive Neuromuscular Facilitation in Shoulder Dysfunction Post Mastectomy
Brief Title: Pilates Exercise Versus Proprioceptive Neuromuscular Facilitation in Shoulder Dysfunction Post Mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Raafat Ahmed Ali, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ahmed-005293
Record Dates: First submitted 2024-10-20; First posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Pilates; Proprioceptive Neuromuscular Fascilitation; Shoulder Dysfunction; Mastectomy
MeSH Terms: interventions — Exercise Movement Techniques; Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pilates exercise (Experimental): This group includes 20 patients who had mastectomy and will recieve Pilates exercise in addition to conventional physical therapy program (stretching exercises and strengthening exercises), and routine medical treatment. Patients will receive 3 sessions per week for 12 weeks, time of session is 45 - 60 min according to patient ability
  Interventions: Other: Pilates exercises
- proprioceptive neuromuscular facilitation (PNF) (Active Comparator): This group includes 20 patients who had mastectomy and will receive PNF exercise in addition to conventional physical therapy program (stretching exercises and strengthening exercises) and routine medical treatment. Patients will receive 3 sessions per week for 12 weeks, time of session is 45 - 60 min according to patient ability
  Interventions: Other: proprioceptive neuromuscular facilitation
- Conventional exercise (Active Comparator): This group includes 20 patients who had mastectomy and will receive conventional physical therapy program (stretching exercises and strengthening exercises) and routine medical treatment. Patients will receive 3 sessions per week for 12 weeks, time of session is 45 - 60 min according to patient ability
  Interventions: Other: The conventional program

INTERVENTIONS:
Other: Pilates exercises — Before starting the training program, patients will learn key Pilates elements, including diaphragmatic breathing, neutral position, rib cage placement, shoulder placement, and head and neck placement. The exercise program includes Pilates-based mat exercises and Pilates-based theraband exercises, with patients placed in supine, prone, and kneeling positions to perform exercises for the affected shoulder. The patient will be placed in various positions for optimal results.
  Arms: Pilates exercise
Other: proprioceptive neuromuscular facilitation — Before starting the training program, patients will learn key Pilates elements, including diaphragmatic breathing, neutral position, rib cage placement, shoulder placement, and head and neck placement. The exercise program includes Pilates-based mat exercises and Pilates-based theraband exercises, with patients placed in supine, prone, and kneeling positions to perform exercises for the affected shoulder. The patient will be placed in various positions for optimal results.
  Arms: proprioceptive neuromuscular facilitation (PNF)
Other: The conventional program — Each patient was in the supine position and will receive stretching exercise for the flexors and adductors, and strengthening for the extensors, abductors and scapular stabilizers of the affected shoulder
  Arms: Conventional exercise

SUMMARY:
The purpose of the study was done to evaluate the therapeutic efficacy of Pilates versus PNF in treatment of shoulder dysfunction and limitation of range of motion after mastectomy

DETAILED DESCRIPTION:
Mastectomy is the removal of the entire breast, with five types: simple or total mastectomy, modified radical mastectomy, radical mastectomy, partial mastectomy, and subcutaneous (nipple-sparing) mastectomy. Post-surgical pain and changes in breast shape can lead to side effects like wound infection, hematoma, seroma, shoulder pain, edema, and decreased range of motion. Mastectomy rates vary worldwide, with the highest rate in central and eastern Europe at 77%. Some women at high risk of breast cancer choose to have a mastectomy even when there's no sign of cancer.

Pilates improve flexibility, build strength, and develop control and endurance in the entire body. It emphasizes alignment, breathing, developing a strong core, and improving coordination and balance. The core, consisting of muscles of the abdomen, low back, and hips, is often called the "powerhouse" and is thought to be the key to a person's stability.

Proprioceptive Neuromuscular Facilitation (PNF) is a stretching technique used to improve muscle elasticity and has been shown to have a positive effect on active and passive range of motions.

ELIGIBILITY:
Inclusion Criteria:

Age range between 40-75 years.

* Only females will participate in the study.
* All patients have no diabetes or blood problems.
* All patients enrolled to the study will have their informed consent

Exclusion Criteria:

Age less than 40 or more than 75 years.

* Diabetes mellitus.
* Subjects suffering from active malignant tumors.
* Subjects treated with skin graft.
* Subjects with Mental illness.
* Subjects with skin diseases
* Subjects with any previous cause for shoulder dysfunction

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — All females who have no diabetes or blood problems.
Enrollment: 60 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
assessment of the change of shoulder range of motion using Software/Smartphone-based Goniometer | at baseline and 3 months
  Smartphones can be used as digital goniometers, offering benefits like convenience, ease of measurement, application-based tracking, and one-hand use. These applications use accelerometers to calculate joint angles. Patients with muscle issues, such as abduction and flexion, may experience reduced range of movement due to muscle bulk loss and bony leverage. However, these patients can compensate with the opposite arm, reducing the impact on daily activities.

SECONDARY OUTCOMES:
Composite assessment of pain and disability using Shoulder pain and disability index | at baseline and 3 months
  It i used to determine the shoulder pain and disability. It comprises of 13 items: a 5-item subscale to evaluate the pain and an 8-item subscale to evaluate the disability. The total score is determined by averaging the pain and disability subscale scores.
  It exhibits great construct validity, associating admirably with other district explicit shoulder questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- out-patient clinic, faculty of physical therapy, Cairo university, Giza, Egypt